CLINICAL TRIAL: NCT04663126
Title: Pilot Study to Test the Feasibility of IV Injected Tc-99m-tilmanocept for Imaging of M2-like Tumour Associated Macrophages in Metastatic Melanoma
Brief Title: Feasibility of IV Tc-99m-tilmanocept for Imaging of M2-like TAMs in Metastatic Melanoma
Acronym: Tilmanocept
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: after inclusion of 5 patients, tracer had low uptake (kidney/liver)
Sponsor: John O. Prior (Other)
Responsible Party: Sponsor-Investigator, John O. Prior, Head of Department, Service of Nuclear Medicine and Molecular Imaging, University of Lausanne Hospitals
Organization: University of Lausanne Hospitals (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Tilmanocept
Record Dates: First submitted 2020-11-30; First posted 2020-12-10 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: Melanoma
Keywords: Macrophages M2
MeSH Terms: conditions — Melanoma | interventions — technetium-diethylenetriaminepentaacetic acid-mannosyl-dextran

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment group (Experimental): Patients diagnosed with advanced melanoma (stage III-IV) will receive IV 250 µg Tilmanocept, labelled with 370 MBq of Tc-99m before the first cycle of clinically scheduled anti-PD-1 immunotherapy.
  Interventions: Drug: Tc-99m tilmanocept

INTERVENTIONS:
Drug: Tc-99m tilmanocept — IV 250 µg Tilmanocept, labelled with 370 MBq of Tc-99m
  Other Names: Lymphoseek

SUMMARY:
This study in 20 patients is designed as a monocentric, open-label and uncontrolled, exploratory pilot study. Patients diagnosed with advanced melanoma (stage III-IV) and scheduled for anti-PD-1 immunotherapy will be recruited for this project. Patients will receive IV 250 µg Tilmanocept, labelled with 370 MBq of Tc-99m (bolus injection) according to the Navidea's protocol in our GMP certified radiopharmaceutical unit, before the first cycle of clinically scheduled immunotherapy.

Scintigraphy images will be acquired dynamically from time of injection to +30 minutes. Quantitative SPECT/CT (xSPECT/CT, Siemens Symbia Intevo, Erlangen, Germany) imaging will be performed up to 1 hour p.i. to evaluate hyperaemia, and up to 3 hours p.i. to image and measure the CD206 receptor uptake. The data of the scans will be compared to immunohistochemistry results from biopsy staining for TAMs and M2-like TAMs and retrospectively with response to the immunotherapy to determine any correlation between M2-like TAMs and treatment response. For the planned retrospective comparison we will use the FDG - PET/CT data that is done after the immunotherapy as standard of care. We will analyse the lesion size and FDG - uptake in standard of care PET/CT of CD206+ and CD206 negative lesions in Tilmanocept SPECT/CT before and after immunotherapy to determine any correlation between CD206 related uptake and treatment response.

DETAILED DESCRIPTION:
According to the Swiss Federal Statistical Office, cancer has been the leading cause of death in Switzerland for men aged between 45 and 84 and women aged between 25 and 84. Melanoma, represents the deadliest and most aggressive form of skin cancer. The incidence of melanoma is rising and in Switzerland it is the fourth most occurring malignancy. In the recent years many advances have been achieved in the treatment of disseminated disease, namely targeted and immunomodulatory treatments (checkpoint inhibitors), either as monotherapy or in combination. Immune checkpoint inhibitors, such as anti-PD-1 are standard of care for advanced melanoma.

However, despite all the success by checkpoint inhibitors, still many patients do not benefit from treatment. Therefore, several attempts have been made to investigate possible prediction of outcome to PD1/PD-L1 treatment. Scientific studies reported mutational load, neoantigens or PD1/PD-L1 expression and/or CD8 infiltrates in melanoma to be predictive for response. However, it has further been shown that also PD-L1 negative tumours respond to PD1/PD-L1 blockade. One possible explanation could be the heterogeneity of intra-tumoural PD-L1 expression or the heterogeneity among different tumour sites in melanoma patients. Overall, the PD-L1 expression is highly dependent on extrinsic factors, as for example hypoxia and therefore highly versatile at different sites and over time.

Another important mechanism of resistance lies in the tumour microenvironment, mainly in inhibitory immune cells of the host. Among others, such as regulatory t-cells (Tregs) or myeloid derived stem cells (MDSC), tumour associated macrophages (TAMs) seem of particular importance in the immune-modulation of the tumour microenvironment.

TAMs in the tumour microenvironment play an essential role in cancer progression. Particularly, the alternatively activated M2 polarized phenotype (M2-like) is confirmed as indicator of poor patients' outcome. During melanoma progression the anti-tumoural M1 polarized phenotype (M1-like) shifts towards the M2 phenotype, which can directly suppress immunity for example via production of cytokines as TGFb or IL-10, cooperating in the reduction of specific CD8 derived immune response. The evolution in understanding the macrophage compartment led therefore to the development of further treatment strategies as CSFR-1 directed antibodies, showing promising synergizing effects with PD-1 directed treatment and reversed resistance to checkpoint inhibitor treatment.

CD206, also termed as MRC1 (C-type mannose receptor 1), is an M2-like macrophage marker in both mouse and human. Its upregulation in macrophages renders them to produce IL-10 and TGFb, identifying this TAM population as anti-inflammatory subtype.

Tc-99m-tilmanocept is a FDA/EMA approved drug (Lymphoseek™, NAVIDEA Biopharmaceuticals, OH, USA). The radio-peptide targets CD206 with nano-molar affinities and is licensed for mapping and localization of lymph nodes draining breast cancer or melanoma using subcutaneous, intradermal, subareolar, or peritumoral injection. Studies have shown superiority to conventional sentinel node procedures. Technetium Tc-99m binds to the diethylenetriaminepentaacetic acid (DTPA) moieties of the Tilmanocept, making it a tracer, suitable for lymph node scintigraphy/SPECT/CT.

Furthermore, recent evidence establishes its role to detect systemic inflammation. Due to its high specificity, even small targets as atherosclerotic plaques in mice can be visualized. Most recent trials have investigated Tc-99m Tilmanocept as intravenous injection (IV) in patients with Rheumatoid Arthritis. A dosage of 150 µg Tilmanocept IV, labelled with 370 MBq of Tc-99m-has demonstrated to be safe and was specific in affected joints of all subjects who had undergone multiple RA flares, which demonstrates CD206+ macrophage infiltration of these joints. Several trials currently investigate the role of Tc-99m-tilmanocept IV and show promising results, for example in patients with Kaposi Sarcoma (NCT03157167) or in patients with liver metastases (NCT03029988).

This study aims to investigate the feasibility and efficacy of Tc-99m-tilmanocept as a marker for CD206+ M2-like TAMs in lesions in melanoma patients. The identification of a correlation of M2-like TAMs presence with the outcome of patients receiving anti-PD1 immunotherapy, would open up new ways to predict ICH treatment response. Therefore, we want to take the first step with this pilot study to evaluate the feasibility of Tc-99m-tilmanocept as a marker for imaging of M2-like TAMs in melanoma metastasis.

This Project falls under risk category C. Intravenous Injection had been tested in a Phase I dose escalation trial in subjects with active rheumatoid arthritis. Subjects received an IV injection of 50, 200 or 400µg Tilmanocept labelled with 37, 185 or 370 MBq of Tc-99m. This study reported that IV injection of Tc-99m-tilmanocept was well tolerated and no adverse drug reactions were observed in any group. Nevertheless, the approval for Tilmanocept does not include IV as route of administration. Therefore, the risk category is C.

There are no data available determining the risk for pregnant woman or the foetus. But, as for every nuclear medicine exam, pregnancy will be tested before any intervention and is part of the standard of care precaution. Pregnancy is an exclusion criterion.

Although no serious hypersensitivity reactions were reported in clinical trials with Tc-99m-tilmanocept, there might be a risk of such reaction due to its chemical similarity to dextran. Patients will be ask before administration about previous hypersensitivity reactions to dextran and modified forms of dextran. In case of emergency, standard emergency procedures will be employed.

There is no immediate benefit to the study participants. The results of the study might provide a better understanding of the diversity of responses to immunotherapy and might allow in future to predict the response of a melanoma patient to immunotherapy. This prediction could allow a more personalized treatment plan for future melanoma patients and could therefore also prevent unnecessary toxicity reactions caused by immunotherapy.

General study design This study in 20 patients is designed as a monocentric, open-label and uncontrolled, exploratory pilot study. Patients diagnosed with advanced melanoma (stage III-IV) and scheduled for anti-PD-1 immunotherapy will be recruited for this project. Patients will receive IV 250 µg Tilmanocept, labelled with 370 MBq of Tc-99m (bolus injection) according to the Navidea's protocol in our GMP certified radiopharmaceutical unit, before the first cycle of clinically scheduled immunotherapy.

Scintigraphy images will be acquired dynamically from time of injection to +30 minutes. Quantitative SPECT/CT (xSPECT/CT, Siemens Symbia Intevo, Erlangen, Germany) imaging will be performed up to 1 hour p.i. to evaluate hyperaemia, and up to 3 hours p.i. to image and measure the CD206 receptor uptake. The data of the scans will be compared to immunohistochemistry results from biopsy staining for TAMs and M2-like TAMs and retrospectively with response to the immunotherapy to determine any correlation between M2-like TAMs and treatment response. For the planned retrospective comparison we will use the FDG - PET/CT data that is done after the immunotherapy as standard of care. We will analyse the lesion size and FDG - uptake in standard of care PET/CT of CD206+ and CD206 negative lesions in Tilmanocept SPECT/CT before and after immunotherapy to determine any correlation between CD206 related uptake and treatment response.

ELIGIBILITY:
Inclusion Criteria:

* Female and male
* Age ≥ 18
* Diagnosis of having advanced melanoma , stage III-IV
* Scheduled for clinically indicated anti-PD-1 immunotherapy
* Informed Consent as documented by signature
* FDG PET/CT within 4 weeks before screening
* Biopsy available
* Minimum 3 lesions detected in FDG PET/CT

Exclusion Criteria:

* Age under 18
* Ocular melanoma
* Women who are pregnant or breast feeding,
* Intention to become pregnant during the course of the study,
* Previous enrolment into the current study,
* Enrolment of the investigator, his/her family members, employees and other dependent persons,
* Previous immunotherapy,
* History of any disease or relevant physical or psychiatric condition or abnormal physical finding which may interfere with the study objectives at the investigator judgment
* The subject has a known allergy to or has had an adverse reaction to dextran exposure
* Insufficient knowledge of project language, inability to give consent or to follow procedures
* The patient makes use of his/her "right not to know" and refuses to be informed about incidental findings

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2023-01-08 (Actual); Study Completion 2023-06-19 (Actual)

PRIMARY OUTCOMES:
Imaging results | 3 hours post injection
  The primary endpoint is the imaging result obtained by scintigraphy/SPECT at day 0 as lesion number and site, compared to standard of care clinical imaging (FDG - PET/CT) per lesion and per patient.

SECONDARY OUTCOMES:
Immunohistochemistry | 1 week after scan
  Secondary endpoint will be the proportion of macrophages and the ratio of macrophage subtype (CD206 positive (M2-like) versus CD206 negative (M1-like)), obtained by immunohistochemistry in biopsies in correlation with Tc-99m-tilmanocept uptake.
Retrospective analysis | 1 week after scan
  For retrospective analysis of correlation of M2-like TAM proportion and response to anti-PD1 immunotherapy we will compare the three most active lesions (uptake of Tc-99m-tilmanocept) in scintigraphy/SPECT images with SOC follow up imaging PET/CT (or if needed other anatomical imaging as MRI or contrast enhanced CT) in each patient.

CONTACTS AND LOCATIONS:
Overall Officials: Niklaus Schaefer, Prof., Principal Investigator — CHUV Lausanne
Locations (1):
- Centre Hospitalier Universitaire Vaudois, Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Domingues B, Lopes JM, Soares P, Populo H. Melanoma treatment in review. Immunotargets Ther. 2018 Jun 7;7:35-49. doi: 10.2147/ITT.S134842. eCollection 2018. PMID 29922629
- [Background] Hodi FS, O'Day SJ, McDermott DF, Weber RW, Sosman JA, Haanen JB, Gonzalez R, Robert C, Schadendorf D, Hassel JC, Akerley W, van den Eertwegh AJ, Lutzky J, Lorigan P, Vaubel JM, Linette GP, Hogg D, Ottensmeier CH, Lebbe C, Peschel C, Quirt I, Clark JI, Wolchok JD, Weber JS, Tian J, Yellin MJ, Nichol GM, Hoos A, Urba WJ. Improved survival with ipilimumab in patients with metastatic melanoma. N Engl J Med. 2010 Aug 19;363(8):711-23. doi: 10.1056/NEJMoa1003466. Epub 2010 Jun 5. PMID 20525992
- [Background] Robert C, Long GV, Brady B, Dutriaux C, Maio M, Mortier L, Hassel JC, Rutkowski P, McNeil C, Kalinka-Warzocha E, Savage KJ, Hernberg MM, Lebbe C, Charles J, Mihalcioiu C, Chiarion-Sileni V, Mauch C, Cognetti F, Arance A, Schmidt H, Schadendorf D, Gogas H, Lundgren-Eriksson L, Horak C, Sharkey B, Waxman IM, Atkinson V, Ascierto PA. Nivolumab in previously untreated melanoma without BRAF mutation. N Engl J Med. 2015 Jan 22;372(4):320-30. doi: 10.1056/NEJMoa1412082. Epub 2014 Nov 16. PMID 25399552
- [Background] Ribas A, Puzanov I, Dummer R, Schadendorf D, Hamid O, Robert C, Hodi FS, Schachter J, Pavlick AC, Lewis KD, Cranmer LD, Blank CU, O'Day SJ, Ascierto PA, Salama AK, Margolin KA, Loquai C, Eigentler TK, Gangadhar TC, Carlino MS, Agarwala SS, Moschos SJ, Sosman JA, Goldinger SM, Shapira-Frommer R, Gonzalez R, Kirkwood JM, Wolchok JD, Eggermont A, Li XN, Zhou W, Zernhelt AM, Lis J, Ebbinghaus S, Kang SP, Daud A. Pembrolizumab versus investigator-choice chemotherapy for ipilimumab-refractory melanoma (KEYNOTE-002): a randomised, controlled, phase 2 trial. Lancet Oncol. 2015 Aug;16(8):908-18. doi: 10.1016/S1470-2045(15)00083-2. Epub 2015 Jun 23. PMID 26115796
- [Background] Larkin J, Chiarion-Sileni V, Gonzalez R, Grob JJ, Cowey CL, Lao CD, Schadendorf D, Dummer R, Smylie M, Rutkowski P, Ferrucci PF, Hill A, Wagstaff J, Carlino MS, Haanen JB, Maio M, Marquez-Rodas I, McArthur GA, Ascierto PA, Long GV, Callahan MK, Postow MA, Grossmann K, Sznol M, Dreno B, Bastholt L, Yang A, Rollin LM, Horak C, Hodi FS, Wolchok JD. Combined Nivolumab and Ipilimumab or Monotherapy in Untreated Melanoma. N Engl J Med. 2015 Jul 2;373(1):23-34. doi: 10.1056/NEJMoa1504030. Epub 2015 May 31. PMID 26027431
- [Background] Snyder A, Makarov V, Merghoub T, Yuan J, Zaretsky JM, Desrichard A, Walsh LA, Postow MA, Wong P, Ho TS, Hollmann TJ, Bruggeman C, Kannan K, Li Y, Elipenahli C, Liu C, Harbison CT, Wang L, Ribas A, Wolchok JD, Chan TA. Genetic basis for clinical response to CTLA-4 blockade in melanoma. N Engl J Med. 2014 Dec 4;371(23):2189-2199. doi: 10.1056/NEJMoa1406498. Epub 2014 Nov 19. PMID 25409260
- [Background] McGranahan N, Furness AJ, Rosenthal R, Ramskov S, Lyngaa R, Saini SK, Jamal-Hanjani M, Wilson GA, Birkbak NJ, Hiley CT, Watkins TB, Shafi S, Murugaesu N, Mitter R, Akarca AU, Linares J, Marafioti T, Henry JY, Van Allen EM, Miao D, Schilling B, Schadendorf D, Garraway LA, Makarov V, Rizvi NA, Snyder A, Hellmann MD, Merghoub T, Wolchok JD, Shukla SA, Wu CJ, Peggs KS, Chan TA, Hadrup SR, Quezada SA, Swanton C. Clonal neoantigens elicit T cell immunoreactivity and sensitivity to immune checkpoint blockade. Science. 2016 Mar 25;351(6280):1463-9. doi: 10.1126/science.aaf1490. Epub 2016 Mar 3. PMID 26940869
- [Background] Tumeh PC, Harview CL, Yearley JH, Shintaku IP, Taylor EJ, Robert L, Chmielowski B, Spasic M, Henry G, Ciobanu V, West AN, Carmona M, Kivork C, Seja E, Cherry G, Gutierrez AJ, Grogan TR, Mateus C, Tomasic G, Glaspy JA, Emerson RO, Robins H, Pierce RH, Elashoff DA, Robert C, Ribas A. PD-1 blockade induces responses by inhibiting adaptive immune resistance. Nature. 2014 Nov 27;515(7528):568-71. doi: 10.1038/nature13954. PMID 25428505
- [Background] Sznol M, Chen L. Antagonist antibodies to PD-1 and B7-H1 (PD-L1) in the treatment of advanced human cancer. Clin Cancer Res. 2013 Mar 1;19(5):1021-34. doi: 10.1158/1078-0432.CCR-12-2063. PMID 23460533
- [Background] Wolchok JD, Kluger H, Callahan MK, Postow MA, Rizvi NA, Lesokhin AM, Segal NH, Ariyan CE, Gordon RA, Reed K, Burke MM, Caldwell A, Kronenberg SA, Agunwamba BU, Zhang X, Lowy I, Inzunza HD, Feely W, Horak CE, Hong Q, Korman AJ, Wigginton JM, Gupta A, Sznol M. Nivolumab plus ipilimumab in advanced melanoma. N Engl J Med. 2013 Jul 11;369(2):122-33. doi: 10.1056/NEJMoa1302369. Epub 2013 Jun 2. PMID 23724867
- [Background] Obeid JM, Erdag G, Smolkin ME, Deacon DH, Patterson JW, Chen L, Bullock TN, Slingluff CL. PD-L1, PD-L2 and PD-1 expression in metastatic melanoma: Correlation with tumor-infiltrating immune cells and clinical outcome. Oncoimmunology. 2016 Sep 20;5(11):e1235107. doi: 10.1080/2162402X.2016.1235107. eCollection 2016. PMID 27999753
- [Background] Madore J, Vilain RE, Menzies AM, Kakavand H, Wilmott JS, Hyman J, Yearley JH, Kefford RF, Thompson JF, Long GV, Hersey P, Scolyer RA. PD-L1 expression in melanoma shows marked heterogeneity within and between patients: implications for anti-PD-1/PD-L1 clinical trials. Pigment Cell Melanoma Res. 2015 May;28(3):245-53. doi: 10.1111/pcmr.12340. Epub 2014 Dec 22. PMID 25477049
- [Background] Barsoum IB, Smallwood CA, Siemens DR, Graham CH. A mechanism of hypoxia-mediated escape from adaptive immunity in cancer cells. Cancer Res. 2014 Feb 1;74(3):665-74. doi: 10.1158/0008-5472.CAN-13-0992. Epub 2013 Dec 13. PMID 24336068
- [Background] Sharma P, Hu-Lieskovan S, Wargo JA, Ribas A. Primary, Adaptive, and Acquired Resistance to Cancer Immunotherapy. Cell. 2017 Feb 9;168(4):707-723. doi: 10.1016/j.cell.2017.01.017. PMID 28187290
- [Background] Siveen KS, Kuttan G. Role of macrophages in tumour progression. Immunol Lett. 2009 Apr 27;123(2):97-102. doi: 10.1016/j.imlet.2009.02.011. Epub 2009 Mar 9. PMID 19428556
- [Background] Falleni M, Savi F, Tosi D, Agape E, Cerri A, Moneghini L, Bulfamante GP. M1 and M2 macrophages' clinicopathological significance in cutaneous melanoma. Melanoma Res. 2017 Jun;27(3):200-210. doi: 10.1097/CMR.0000000000000352. PMID 28272106
- [Background] Qian BZ, Pollard JW. Macrophage diversity enhances tumor progression and metastasis. Cell. 2010 Apr 2;141(1):39-51. doi: 10.1016/j.cell.2010.03.014. PMID 20371344
- [Background] Sun Z, Fourcade J, Pagliano O, Chauvin JM, Sander C, Kirkwood JM, Zarour HM. IL10 and PD-1 Cooperate to Limit the Activity of Tumor-Specific CD8+ T Cells. Cancer Res. 2015 Apr 15;75(8):1635-44. doi: 10.1158/0008-5472.CAN-14-3016. Epub 2015 Feb 26. PMID 25720800
- [Background] Cannarile MA, Weisser M, Jacob W, Jegg AM, Ries CH, Ruttinger D. Colony-stimulating factor 1 receptor (CSF1R) inhibitors in cancer therapy. J Immunother Cancer. 2017 Jul 18;5(1):53. doi: 10.1186/s40425-017-0257-y. PMID 28716061
- [Background] Zhu Y, Knolhoff BL, Meyer MA, Nywening TM, West BL, Luo J, Wang-Gillam A, Goedegebuure SP, Linehan DC, DeNardo DG. CSF1/CSF1R blockade reprograms tumor-infiltrating macrophages and improves response to T-cell checkpoint immunotherapy in pancreatic cancer models. Cancer Res. 2014 Sep 15;74(18):5057-69. doi: 10.1158/0008-5472.CAN-13-3723. Epub 2014 Jul 31. PMID 25082815
- [Background] Stein M, Keshav S, Harris N, Gordon S. Interleukin 4 potently enhances murine macrophage mannose receptor activity: a marker of alternative immunologic macrophage activation. J Exp Med. 1992 Jul 1;176(1):287-92. doi: 10.1084/jem.176.1.287. PMID 1613462
- [Background] Porcheray F, Viaud S, Rimaniol AC, Leone C, Samah B, Dereuddre-Bosquet N, Dormont D, Gras G. Macrophage activation switching: an asset for the resolution of inflammation. Clin Exp Immunol. 2005 Dec;142(3):481-9. doi: 10.1111/j.1365-2249.2005.02934.x. PMID 16297160
- [Background] Bellon T, Martinez V, Lucendo B, del Peso G, Castro MJ, Aroeira LS, Rodriguez-Sanz A, Ossorio M, Sanchez-Villanueva R, Selgas R, Bajo MA. Alternative activation of macrophages in human peritoneum: implications for peritoneal fibrosis. Nephrol Dial Transplant. 2011 Sep;26(9):2995-3005. doi: 10.1093/ndt/gfq771. Epub 2011 Feb 15. PMID 21324976
- [Background] Svensson-Arvelund J, Mehta RB, Lindau R, Mirrasekhian E, Rodriguez-Martinez H, Berg G, Lash GE, Jenmalm MC, Ernerudh J. The human fetal placenta promotes tolerance against the semiallogeneic fetus by inducing regulatory T cells and homeostatic M2 macrophages. J Immunol. 2015 Feb 15;194(4):1534-44. doi: 10.4049/jimmunol.1401536. Epub 2015 Jan 5. PMID 25560409
- [Background] Wallace AM, Han LK, Povoski SP, Deck K, Schneebaum S, Hall NC, Hoh CK, Limmer KK, Krontiras H, Frazier TG, Cox C, Avisar E, Faries M, King DW, Christman L, Vera DR. Comparative evaluation of [(99m)tc]tilmanocept for sentinel lymph node mapping in breast cancer patients: results of two phase 3 trials. Ann Surg Oncol. 2013 Aug;20(8):2590-9. doi: 10.1245/s10434-013-2887-8. Epub 2013 Mar 17. PMID 23504141
- [Background] Baker JL, Pu M, Tokin CA, Hoh CK, Vera DR, Messer K, Wallace AM. Comparison of [(99m)Tc]tilmanocept and filtered [(99m)Tc]sulfur colloid for identification of SLNs in breast cancer patients. Ann Surg Oncol. 2015 Jan;22(1):40-5. doi: 10.1245/s10434-014-3892-2. Epub 2014 Jul 29. PMID 25069859
- [Background] Azad AK, Rajaram MV, Metz WL, Cope FO, Blue MS, Vera DR, Schlesinger LS. gamma-Tilmanocept, a New Radiopharmaceutical Tracer for Cancer Sentinel Lymph Nodes, Binds to the Mannose Receptor (CD206). J Immunol. 2015 Sep 1;195(5):2019-29. doi: 10.4049/jimmunol.1402005. Epub 2015 Jul 22. PMID 26202986
- [Background] Varasteh Z, Hyafil F, Anizan N, Diallo D, Aid-Launais R, Mohanta S, Li Y, Braeuer M, Steiger K, Vigne J, Qin Z, Nekolla SG, Fabre JE, Doring Y, Le Guludec D, Habenicht A, Vera DR, Schwaiger M. Targeting mannose receptor expression on macrophages in atherosclerotic plaques of apolipoprotein E-knockout mice using 111In-tilmanocept. EJNMMI Res. 2017 Dec;7(1):40. doi: 10.1186/s13550-017-0287-y. Epub 2017 May 3. PMID 28470406
- [Background] Kardan A, A.B., Sanders J, Kissling A, Ralph D, Shuping J, Blue M, Hartings C, Hershey R, Ismail A, Gierach I, Bailey H, Spaulding A, Haynam M, Zubal G, Cope F., Evaluation of Intravenous Injection of Tc 99m Tilmanocept in Static Planar Gamma Emission Imaging and Fused SPECT/CT Imaging for Rheumatoid Arthritis [abstract]. Arthritis Rheumatol. , 2017. 69.
- [Background] Julious, S.A., Sample size of 12 per group rule of thumb for a pilot study. Pharmaceutical Statistics, 2005. 4(4): p. 287-291.
- [Background] Browne RH. On the use of a pilot sample for sample size determination. Stat Med. 1995 Sep 15;14(17):1933-40. doi: 10.1002/sim.4780141709. PMID 8532986
- [Background] Kardan, A., et al., Intravenous 99mTc-tilmanocept in Planar and Fused SPECT/CT Imaging of Activated Macrophage Infiltration in Subjects with Active Rheumatoid Arthritis. Vol. 59. 2018.
- [Derived] Boughdad S, Latifyan S, Schottelius M, Blue M, Tissot S, Geldhof C, Costes J, Prior JO, Schaefer N. Utility of [99mTc]Tc-tilmanocept, an immunosuppressive macrophage functional imaging agent in melanoma patients receiving checkpoint inhibitor treatment: a feasibility study. Cancer Immunol Immunother. 2025 Sep 6;74(10):298. doi: 10.1007/s00262-025-04127-8. PMID 40913745